CLINICAL TRIAL: NCT05196971
Title: A Phase Ib，Randomized, Double-Blind, Placebo-Controlled Study Evaluating The Safety, Tolerability And Pharmacokinetics of HS-10345 In Chinese Adult Subjects With Treatment Resistant Depression
Brief Title: A Study To Evaluate The Safety, Tolerability And Pharmacokinetics of HS-10345 In Treatment-Resistant Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10345-102
Record Dates: First submitted 2022-01-09; First posted 2022-01-19 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Treatment Resistant Depressive Disorder
Keywords: Treatment resistant depressive disorder; Intranasal; HS-10345
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10345 84mg (Experimental): Participants will self-administer intranasal HS-10345 84mg on Days 1, 4, 8, and 11 during the double-blind phase
  Interventions: Drug: HS-10345 84mg
- Placebo (Placebo Comparator): Participants will be self-administered on Days 1, 4, 8, and 11 during the double-blind phase
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10345 84mg — 6 sprays of HS-10345 84 mg self-administered as an intranasal formulation for 4 days (Days 1, 4, 8, 11) during the double-blind phase
  Other Names: HS-10345
  Arms: HS-10345 84mg
Drug: Placebo — 6 sprays of placebo self-administered as an intranasal formulation for 4 days (Days 1, 4, 8, 11) during the double-blind phase
  Other Names: HS-10345 Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of intranasal HS-10345 (84mg) compared with placebo in participants with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, multicenter study. Approximately 24 male and female adult participants diagnosed with TRD will participant in this study. There will be 4 study phases: a 4-week screening phase, a 1-day baseline phase, a double-blind treatment phase (Day 1 to Day 15), and a 1-week post-treatment (follow-up) phase. Firstly, 12 patients will be assigned to intranasal placebo or HS-10345 of 84mg. Extra 12 patients may be enrolled depending on the pharmacokinetics analysis of 84mg. Safety assessments will be performed throughout the study. The maximum study duration for a participant will be 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
2. Participant must meet Diagnostic and Statistical Manual of Mental Disorders -5 Edition -Text Revised (DSM-5) diagnostic criteria for Major Depressive Disorder (MDD), without psychotic features, based upon clinical assessment, and confirmed by the Mini International Neuropsychiatric Interview (MINI).
3. Participant must have had an inadequate response to at least 1 antidepressants in the current episode of depression assessed by the antidepressant treatment response questionnaire (ATRQ), and was taking another oral antidepressant 2 weeks before entering the screening period which will be assessed "non-response" by Montgomery Asberg Depression Rating Scale (MADRS) during the screening period, defined as MADRS total score reduced ≤25%.
4. Comfortable with self-administration of intranasal medication and able to follow instructions provided.
5. A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) at Screening and a negative urine pregnancy test prior to Period 1 randomization on Day 1.

Exclusion Criteria:

1. Subject has a current DSM-5 diagnosis of psychotic disorder, MDD with psychosis, bipolar, obsessive compulsive disorder (OCD), intellectual disability, Autism spectrum Disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, and narcissistic personality disorder.
2. Subject has suicidal ideation with intent to act within the past 6 months based on the Columbia-Suicide Severity Rating Scale (C-SSRS), or has a history of suicidal behavior within the past year as assessed on the C-SSRS.
3. Subject has uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg) despite diet, exercise or a stable dose of a permitted anti-hypertensive treatment at Screening or Day 1 prior to Period 1 randomization; or any past history of hypertensive crisis.
4. Subject had a history of severe pulmonary insufficiency or SpO2<93% at screening time or prior to dosing.
5. Anatomical or medical conditions that may impede delivery or absorption of study medication.
6. Subject is a woman who is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or within 12 weeks after the last dose of study drug.
7. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody and human immunodeficiency virus (HIV) antibody tests positive.
8. Subject has had major surgery, (e.g., requiring general anesthesia) within 12 weeks before screening, or has surgery planned during the time the subject is expected to participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and Serious Adverse Events (SAEs) | up to 7 weeks
  Participants during hospitalization will be closely observed to assure maximal safety and to collect occurrence of all adverse event. To follow-up on the 7th day after discharge, all participants will return to the hospital for information regarding their health condition. All adverse events will be collected with special attention to occurrence of psychotomimetic and dissociative effects after study drug administration.
Change from Baseline (Day -1) in Columbia-Suicide Severity Rating Scale (C-SSRS) Total Score at Day 15 in the Double-Blind Treatment Phase | up to 15 days
  This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale. A negative change in score indicates improvement.
Change from Baseline (Day -1) in The Clinician Administered Dissociative States Scale (CADSS) Total Score at 40 minutes and 2 hours after dosing in the Double-Blind Treatment Phase- ANCOVA Analysis on Ranks | up to 2 hours
  This scale is intended to be used to assess the dissociative states of participants. It contains 23 objective items, every item ranges from 0 to 4. A negative change in score indicates improvement.
Change From pre-dosing in Modified Observer's Assessment of Alertness and Sedation (MOAA/S) Total Score at 20 minutes、40 minutes and 2 hours after dosing in the Double-Blind Treatment Phase- ANCOVA Analysis on Ranks | up to 2 hours
  The Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scale is frequently used in sedation-related drug and device studies to assess a subject's level of sedation. It ranges from 0 to 5, with a score of 5 defined as awake or minimally sedated, and a score of 0 defined as general anesthesia. This scale is intended to be used by individuals who have received training in its administration. A positive change in score indicates improvement.
Change from Baseline (Day -1) in Physician Withdrawal Checklist (PWC-20) Total Score at Day 15 in the Double-Blind Treatment Phase and Day 21 in the Follow-Up Phase- ANCOVA Analysis on Ranks | up to 15 days
  The PWC-20 was developed to detect any potential BZ-like treatment discontinuation (withdrawal) symptoms caused by experimental anxiolytics of the non-SSRI type. A negative change in score indicates improvement.

SECONDARY OUTCOMES:
Cmax - maximum HS-10345 plasma concentration | up to 72 hours after each study drug administration
  The maximum concentration of the HS-10345 in plasma after drug administration, obtained directly from the measured concentrations.
AUC (0-24) - area under the HS-10345 plasma concentration-time curve from time 0 to 24 hours after study drug administration | up to 24 hours after each study drug administration
  The AUC (0-24) is a measure of total plasma exposure to the drug from time point zero to 24 hours after study drug administration.
Tmax - time to reach maximum HS-10345 plasma concentration | up to 72 hours after each study drug administration
  The Tmax is time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times.
AUC (0-inf) - area under the HS-10345 plasma concentration-time curve from time 0 to infinity time | up to 72 hours after each study drug administration
  The AUC(0-inf) is a measure of total plasma exposure to the drug from time point zero extrapolated to infinity
T1/2 - plasma elimination half-life for HS-10345 | up to 72 hours after each study drug administration
  T1/2 will be calculated as 0.693/Kel
Change from Baseline (Day -1) in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Day 2/8/15- Analysis of Covariance (ANCOVA) Analysis | up to 15 days
  MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. A negative change in score indicates improvement

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality, China